CLINICAL TRIAL: NCT03399201
Title: The Effect of General or Spinal Anesthesia on Pulmonary Function Tests in Geriatric Patients
Brief Title: The Effect of Anesthesia Type on Pulmonary Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, Associate Professor,MD, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Spiro
Record Dates: First submitted 2017-12-22; First posted 2018-01-16 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Anesthesia; Geriatric Patients
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (Active Comparator): Standard General Anesthesia will be applied.The change of the pulmonary functions will be evaluated via spirometer.
  Interventions: Procedure: General anesthesia; Diagnostic Test: Spirometer
- Neuraxial Anesthesia (Active Comparator): Neuraxial anesthesia will be applied. The change of the pulmonary functions will be evaluated via spirometer.
  Interventions: Procedure: Neuraxial anesthesia; Diagnostic Test: Spirometer

INTERVENTIONS:
Procedure: General anesthesia — induction with the intravenous anesthetic (Propofol) and maintenance with the inhalational anesthetic (Sevoflurane)
  Arms: General Anesthesia
Procedure: Neuraxial anesthesia — Spinal anesthesia will be applied via the local anesthetic ( Bupivacaine).
  Arms: Neuraxial Anesthesia
Diagnostic Test: Spirometer — Pulmonary function will be evaluated via the portable spirometer (MIR Spirodoc, Spirodoc®, Roma, Italy)

SUMMARY:
The role of neuraxial anesthesia in preventing respiratory complications is a controversial in elderly patients. The aim of the study was to evaluate the benefits of neuraxial anesthesia on pulmonary function during post-operative term in geriatric patients undergoing to elective non-abdominal surgery.

DETAILED DESCRIPTION:
Sixty elder patients will be randomly assigned to General anesthesia or Neuraxial anesthesia groups. Spirometry, will be performed at pre-operative and post-operative terms. Pulmonary function tests will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age
* Undergoing non-abdominal surgery under anesthesia in supine position

Exclusion Criteria:

* Pulmonary disease
* Hematological disease
* Undergoing Abdominal surgery
* Non-supine position during surgery
* Nicotine Abuse

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
The changes on forced vital capacity | At Preoperative, postoperative 2. hours, postoperative 24. hours
  Forced vital capacity will be measured via spirometer
The changes on forced expiratory volume in 1 s | At Preoperative, postoperative 2. hours, postoperative 24. hours
  Forced expiratory volume in 1 s will be measured via spirometer
The changes on mid-expiratory flow (MEF 25-75) | At Preoperative, postoperative 2. hours, postoperative 24. hours
  mid-expiratory flow (MEF 25-75) will be measured via spirometer
The changes on peak expiratory flow (PEF) | At Preoperative, postoperative 2. hours, postoperative 24. hours
  Peak expiratory flow (PEF) will be measured by the spirometer

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Karaman, MD, Principal Investigator — Associate Professor
Locations (1):
- Gaziosmanpasa University Hospital, Tokat Province, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No